CLINICAL TRIAL: NCT02283073
Title: PDx Biomarker Assay Study for the Diagnosis of Parkinson's Disease
Brief Title: Study for the Early Diagnosis of Parkinson's Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Bio Shai Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: PDx001; 82/14 (Other: Assaf HaRofeh); TASMC -14-TG-0489-14-TLV-CTIL (Other: Tel Aviv Sourasky Medical Center); 1735-14-SMC (Other: Sheba Medical Center); 0463-14-RMB (Other: Rambam Health Care Campus)
Record Dates: First submitted 2014-10-27; First posted 2014-11-05 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Parkinson's Disease, Idiopathic
Keywords: Diagnosis
MeSH Terms: conditions — Parkinson Disease; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The mRNA in blood samples will be transcribed to cDNA.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Idiopathic Parkinson's disease: Patient with clinical diagnosis of Idiopathic Parkinson's Disease according to Queen Square Brain Bank Criteria up to one year prior to enrollment in study.
- Differential Diagnosis Group: MSA, PSP, CBD, Lewy body dementia, Essential Tremor, and Healthy Controls

SUMMARY:
The main objective of the study is to design and validate the blood based PDx gene expression and miRNA assay for the early diagnosis of Parkinson's disease patients. Differential diagnosis includes patients with Multiple System Atrophy, Progressive Supranuclear Palsy, Corticobasal Degeneration, Lewy Body Dementia, Essential Tremor and Normal Controls.

DETAILED DESCRIPTION:
In this study, the PDx assay will be designed and validated in order to distinguish between Idiopathic Parkinson's disease (PD) to patients with similar symptoms and healthy controls. The differential diagnosis cohort includes patients diagnosed with Multiple System Atrophy (MSA), Progressive Supranuclear Palsy (PSP), Corticobasal Degeneration (CBD), Essential Tremor (ET) or Lewy Body Dementia (LBD) and Healthy Controls.

This is a prospective observational study. Blood samples and clinical data will be collected at the first and only study visit. The expression levels of 5 to 6 genes will be analyzed by blinding technicians concerning the diagnosis, demographic data and clinical data, which will be revealed after sending PDx gene expression values to the clinical sites. The gene expression levels will be compared between Parkinson's disease patients to the differential diagnosis cohort and healthy controls. Additional mRNA and miRNA markers will be explored. The primary aim of the study is to design and validate a clinical classifier that will aid the physician in the diagnosis of Parkinson's disease patients. The analysis will be performed in two stages: Stage 1) Exploration analysis and Stage 2) Validation. After one year of taking a blood sample, the study physician will contacted to confirm the patient's diagnosis.

Blood samples will be collected at specialized movement disorder clinics.

Medical history, clinical diagnostic features, family history in regard to Parkinson's disease, use of medication and routine imaging assessment (not mandatory) will be collected at the first and only patient visit.

ELIGIBILITY:
Inclusion Criteria:

* Patient is able and willing to read the informed consent form
* Patient with clinical diagnosis of Idiopathic Parkinson's Disease according to Queen Square Brain Bank Criteria up to one year prior to enrollment in study
* Patient with diagnosis of MSA, PSP, CBD, Lewy Body Dementia, Essential Tremor or Healthy Control
* Men and Women aged 40-80 years
* Willing and able to comply with procurement of blood sample

Exclusion Criteria:

* Any medical, psychiatric or other conditions which, in the opinion of the investigator, would preclude participation
* Pregnancy

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Movement disorder clinics
Sampling Method: Probability Sample
Enrollment: 410 (Actual)
Dates: Start 2014-11; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The Diagnostic Accuracy of PDx mRNA Assay in Diagnosing Idiopathic Parkinson's Disease | One year from enrollment
  Investigate the diagnostic accuracy of the PDx gene expression assay, comprised of 5-6 expressed genes (mRNA - RQ-PCR), to differentiate patients with Idiopathic Parkinson's disease from the Differential Diagnosis Group. Diagnostic Accuracy includes sensitivity, specificity, likelihood ratios and the area under the receiver operating characteristic (ROC) curve. Diagnostic Accuracy will be calculated by comparing the PDx assay results to the Gold Standard Diagnosis, which will be the Clinical diagnosis of the Patient one year after the first and only visit (day of blood collection). The physician investigator will be contacted if there was any change in the baseline diagnosis one year after blood collection according to routine clinical findings.

SECONDARY OUTCOMES:
Diagnostic Accuracy of each one of the PDx assay's expressed genes for Differentiating Idiopathic Parkinson's Disease Patients from Atypical Parkinsonism Patients. | One year from enrollment
  Investigate the diagnostic accuracy (sensitivity, specificity, likelihood ratios and AUC) of each one of the PDx assay expressed genes (RQ-PCR) to differentiate Idiopathic Parkinson's Disease Patients from Atypical Parkinsonism Patients.
Diagnostic Accuracy of each one of the PDx assay's expressed genes for Differentiating Idiopathic Parkinson's Disease Patients from Essential Tremor Patients. | One year from enrollment
  Investigate the diagnostic accuracy (sensitivity, specificity, likelihood ratios and AUC) of each one of the PDx assay expressed genes (RQ-PCR) to differentiate Idiopathic Parkinson's Disease Patients from Essential Tremor Patients.
Diagnostic Accuracy of each one of the PDx assay's expressed genes for Differentiating Idiopathic Parkinson's Disease Patients from Healthy Controls. | One year from enrollment
  Investigate the diagnostic accuracy (sensitivity, specificity, likelihood ratios and AUC) of each one of the PDx assay expressed genes (RQ-PCR) to differentiate Idiopathic Parkinson's Disease Patients from Healthy Controls.

CONTACTS AND LOCATIONS:
Overall Officials: Ofer Gonen, MD, Principal Investigator — Assaf-Harofeh Medical Center
Locations (6):
- Israel (5):
  - Rambam Health Care Campus, Haifa
  - Rabin Medical Center, Petach Tikvah
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Chaim Sheba Medical Center, Tel Litwinsky
  - Assaf Harofeh Medical Center, Ẕerifin
- Pisa University Hospital, Pisa, Italy

REFERENCES:
- [Background] Berardelli A, Wenning GK, Antonini A, Berg D, Bloem BR, Bonifati V, Brooks D, Burn DJ, Colosimo C, Fanciulli A, Ferreira J, Gasser T, Grandas F, Kanovsky P, Kostic V, Kulisevsky J, Oertel W, Poewe W, Reese JP, Relja M, Ruzicka E, Schrag A, Seppi K, Taba P, Vidailhet M. EFNS/MDS-ES/ENS [corrected] recommendations for the diagnosis of Parkinson's disease. Eur J Neurol. 2013 Jan;20(1):16-34. doi: 10.1111/ene.12022. PMID 23279440
- [Derived] Ma YM, Zhao L. Mechanism and Therapeutic Prospect of miRNAs in Neurodegenerative Diseases. Behav Neurol. 2023 Nov 23;2023:8537296. doi: 10.1155/2023/8537296. eCollection 2023. PMID 38058356